CLINICAL TRIAL: NCT02568540
Title: preSmartphone App for Monitoring and Reporting of Hepatitis C Related Health Information: C Tracker Hepatitis C, Care & Collaboration - Patient Reported Outcomes Survey Study
Brief Title: C Tracker, Hepatitis C, Care & Collaboration - Patient Reported Outcomes Survey Study
Acronym: CTracker
Status: Terminated | Type: Observational
Why Stopped: Lack of enrollment
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Kenneth Mandl, Chair in Biomedical Informatics and Population Health and Director, Computational Health informatics Program, Boston Children's Hospital
Other Study IDs: P00018023
Record Dates: First submitted 2015-10-02; First posted 2015-10-06 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; Smartphone; app; Tracker; C Tracker
MeSH Terms: conditions — Hepatitis C; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Today's mobile devices (especially smartphones) are powerful ways to communicate new information to medical researchers. For this study, researchers at Boston Children's Hospital are asking people with hepatitis C to make use of their smartphones to help report information about themselves that may improve how hepatitis C is treated. This study uses a free app called C Tracker that can be installed from the Apple App Store onto the participants iPhone. The main goal of this research study is to use this app to report hepatitis C related health information to the researchers who are conducting this study. The investigators will ask participants about their health,activities, medications, and ways in which hepatitis C has impacted you. This information will be reported anonymously, which means that the researchers doing the study won't know who the participants are.

DETAILED DESCRIPTION:
Specific Aims/Objectives

Aim 1. Develop a free iPhone app ("C TRACKER") designed to anonymously record and report Hepatitis C related health data to study investigators via periodic patient-reported surveys.

Aim 2. Examine the feasibility of enrolling a large cohort of geographically dispersed cohort of subjects with hepatitis C who download and install the C TRACKER app, provide informed consent using the app, and complete study surveys using the app. The app will be made available to the public via the Apple App Store at no cost.

Aim 3. Pilot usage of the app to track and analyze longitudinal measures of hepatitis C related health concerns, physical function, and physical activity via selected disease-specific as well as more broadly applicable patient-reported instruments, including regarding work productivity (WPAI-Hepatitis C), physical functioning (subsets/subscales of the MOS SF-36), physical activity (collected through Apple HealthKit), and prescribed medications.

ELIGIBILITY:
Inclusion Criteria:

* Self-report a diagnosis of Hepatitis C
* English speaking individuals
* 18 years or older
* Must have access to an iPhone that operates on iOS version 8 or higher
* Be able to download apps from the U.S. Apple iPhone Store, and enter data themselves or via a proxy on their behalf

Exclusion Criteria:

• Individuals not meeting inclusion criteria will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who have been diagnosed with Hepatitis C.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2015-10; Primary Completion 2017-12-04 (Actual); Study Completion 2019-01-16 (Actual)

PRIMARY OUTCOMES:
Changes in hepatitis C medication therapy | every 4 months for 2 years
  Patient reported hepatitis C medication therapy. Medication type and timing will be compared against other patient-reported outcome measures looking at workforce productivity and physical health and function. Medication changes will be collected every 4 months (3 times a year).
Changes in Workforce Productivity and Activity Impairment Compared to changes in hepatitis C medication therapy. | every 2 weeks and data will be analyzed every 6 months, for a total of 2 years
  The Work Productivity and Activity Impairment Questionnaire: Hepatitis C V2.0 (WPAI:Hepatitis C, 6 questions in total) will be administered and compared to changes in Hepatitis C medication therapy. Measures will be collected every 2 weeks and data will be analyzed every 6 months.
Changes in Physical Function and Limitations Due to Physical Health Compared to changes in hepatitis C medication therapy. | every 4 months for 2 years; a subset will be analyzed every 2 weeks and data will be analyzed every 6 months, for a total of 2 years
  3. The Physical Function domain and Role Limitations Due to Physical Health domain of the Medical Outcomes Study (MOS) 36-Item Short Form Survey (14 questions in total) will be administered and compared to changes in Hepatitis C medication therapy. All questions will be collected every 4 months. A subset of The Physical Function domain and Role Limitations Due to Physical Health domain of the Medical Outcomes Study (MOS) 36-Item Short Form Survey (5 questions in total) will be administered every 2 weeks. Data will be analyzed every 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States